CLINICAL TRIAL: NCT01343173
Title: Multicenter Trial Estimating the Persistence of Molecular Remission in Chronic Myeloid Leukaemia in Long Term After Stopping Imatinib
Acronym: STIM 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2010/25
Record Dates: First submitted 2011-03-23; First posted 2011-04-27 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Chronic Myeloid Leukaemia
Keywords: Leukemia; Adult Chronic; Myeloid
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients (Experimental)
  Interventions: Drug: Imatinib stop

INTERVENTIONS:
Drug: Imatinib stop — To stop imatinib after inclusion.

SUMMARY:
Background: Complete molecular remission under imatinib, therapeutic interruption possible for patients in complete remission proved in different trials.

Purpose: Stopping imatinib in patients with chronic myeloid leukemia in complete molecular remission during two following years. The objectives of this study are to determine the rate of patients without a molecular relapse and so the rate of molecular relapse, to determine and to seek for clinical and biological CML-related factors predictive for a molecular relapse after imatinib discontinuation. These objectives require to increase the number of study patients to be enrolled for accurate statistical considerations. It will allow to predict which patients have to be proposed for discontinuation without risk of molecular relapse and to select the patients who need to continue or reinforce the treatment to achieve a complete long term eradication of the disease.

DETAILED DESCRIPTION:
The gold standard for the treatment of chronic myeloid leukaemia (CML) is Imatinib, the first tyrosine inhibitor (TKI) of BCR-ABL. Imatinib specifically targets the BCR-ABL tyrosine kinase encoded by the BCR-ABL fusion gene, the molecular hallmark of CML. Regular monitoring of BCR-ABL transcript levels by quantitative RT-PCR is of key importance for the assessment of treatment response to imatinib.

Over time, an increasing proportion of imatinib-treated patients obtain a complete molecular response (CMR), defined as an undetectable molecular residual disease. In a previous study, STIM trial (PHRC 2006, stop Imatinib), 100 patients were included. The preliminary analysis among 69 patients having a median follow up of 21 months shows that the probability to maintain the CMR at 12 months is 45%. Our goal is actually to include up to 200 patients and then let the STIM opened during 3 years in a way to determine the predictive factors of the molecular relapse Discontinuation of treatment is proposed after checking selection criteria and signing informed consent. The assessment of BCR-ABL in peripheral blood by quantitative RT-PCR is performed every month during the first year then every two months second year then every three months during 3 years.

The molecular relapse after imatinib discontinuation is defined by positive PCR for BCR-ABL two times using RTQ-PCR with increasing of the transcript on two following assessment and or a value> 0.1% i.e. lost of MMR. In case of molecular relapse it is recommended to re-challenge an imatinib treatment. According to our experience the 50 patients well documented who re challenged the treatment were sensitive again. The treatment of molecular relapse by second generation tyrosine kinase inhibitors (dasatinib or nilotinib) will possible in the current trial. It is important for all the French patients to be included in a national trial to avoid discontinuation without evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older.
* Chronic myeloid leukaemia in chronic or accelerated phase under treatment with imatinib for at least 3 years.
* Complete molecular remission under treatment with imatinib for at least 2 years.
* HIV serology negative and absence of chronic hepatitis B or C.
* Molecular monitoring according to the international recommendations before the beginning of the study
* For the women old enough to procreate, method of effective contraception
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent.

Exclusion Criteria:

* Under 18 years old.
* Pregnant at the inclusion's time.
* Hospitalized patients without consent.
* Adults under law protection or without ability to assent.
* Previous or planned allogeneic stem cell transplantation.
* HIV serology positive or chronic hepatitis B or C.
* Interfering treatment (corticosteroids, immunosuppressors, chemotherapy, radiotherapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2011-04-06 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Rate of molecular relapse defined by the rate of patients having a significant increasing of BCR-ABL transcript. | Every months during two years

SECONDARY OUTCOMES:
Overall survival | after two years
  Number of patients alive or died will be measured
Clinical and biological profile of patient with complete molecular remission persistence | after two years
  The relevant clinical and biological factors which could be predictive of the the complete molecular remission persistence will be measured by dosage in the blood.
Treatment costs according to days without imatinib. | after two years
Event-free survival | after two years
  All adverse events will be reported to know what kind of adverse events occured to patients without treatment, number of patients with adverse events and in particular number of patients with lost of complete molecular remission.

CONTACTS AND LOCATIONS:
Overall Officials: François-Xavier MAHON, Pr, Principal Investigator — University Hospital Bordeaux, France
Locations (32):
- France (32):
  - University Hospital Angers, Angers
  - CH Annecy, Annecy
  - CHU Bensançon, Besançon
  - Institut Bergonié, Bordeaux
  - Hôpital Morvan, Brest
  - CHU Caen, Caen
  - Hôpitaux civils de Colmar, Colmar
  - CH Sud Francilien, Corbeil-Essonnes
  - Hôpital Henri-Mondor, Créteil
  - CHU Grenoble, Grenoble
  - Centre Hospitalier - La Roche sur Yon, La Roche-sur-Yon
  - Lille University hospital - Hôpital Claude Huriez, Lille
  - CHU Dupuytren, Limoges
  - Hôpital Edouard Herriot, Lyon
  - Institut Paoli Calmette, Marseille
  - CHU Hôtel-Dieu, Nantes
  - Centre Hospitalier de Nevers, Nevers
  - CHU de Nice - Hôpital Archet 1, Nice
  - Hôpital Saint Louis, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - University Hospital Bordeaux, Hôpital du Haut Lévêque, Pessac
  - University Hospital Poitiers - Hôpital Jean Bernard, Poitiers
  - Hôpital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - CH Yves Le Foll, Saint-Brieuc
  - CHR La Réunion, Saint-Denis
  - CH Régional de l'ILE DE LA REUNION/ Groupe Hospitalier Sud, Saint-Pierre
  - Hôpital Purpan, Toulouse
  - CH Valence, Valence
  - C.H.U. Brabois, Vandœuvre-lès-Nancy
  - CH Bretagne Atlantique, Vannes
  - Centre Hospitalier de Versailles - Hôpital André Mignot, Versailles